CLINICAL TRIAL: NCT02336516
Title: Azithromycin in Post Diarrheal Haemolytic and Uremic Syndrome
Acronym: ZITHROSHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P130910 / AOM13540; 2014-001740-38 (EudraCT Number)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Haemolytic and Uremic Syndrome
MeSH Terms: conditions — Hemolysis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin (Experimental): ZITHROMAX ® 40mg/ml solution. DCI : Azithromycin . Pfizer ®
  Interventions: Drug: Azithromycin
- Glucose solution 10% (Placebo Comparator): Glucose solution 10%
  Interventions: Drug: Placebo (glucose solution 10%)

INTERVENTIONS:
Drug: Azithromycin — ZITHROMAX ® 40mg/ml solution. DCI : Azithromycin . Pfizer ® 20mg/kg dose with a maximum dose of 500mg per day for three days
  Arms: Azithromycin
Drug: Placebo (glucose solution 10%)
  Arms: Glucose solution 10%

SUMMARY:
Post diarrheal hemolytic and uremic syndrome (D+HUS) is the first etiology of acute renal failure in children less than 5 years old in France. Previous works highlighted a mortality rate of 2 % and a prevalence of renal sequelae at one year after D+HUS onset in 25 % of patients D+HUS is a consequence of a gastrointestinal infection with shiga toxin (Stx) producing E.coli (STEC). The most frequent straight is E.coli O157H7. The sequence of STEC induced HUS is now well known. Typically, digestive symptoms appear five days following STEC ingestion. STEC colonize the intestinal mucosa, adhere to the enterocyte and cause a typical attaching/effacing lesion and inflammation. Then, diarrhea and vomiting occurred. D+HUS occurs in about 10% of patients and is a consequence of Stx systemic absorption. Indeed, Stx are released in the gastrointestinal tract, then after transferred to the systemic circulation. At the cellular level, Stx binds the globotriosylceramide (Gb3Cer) localized at the surface of the endothelial and epithelial cells of target organs. Following binding to Gb3Cer, the A subunits of Stx are internalized and trigger the activation of the apoptotic program leading to cell death. In addition, Stx are also able to enhance the production and the release of pro inflammatory factor (IL-1, TNFα, IL-6). Cytokines locally produced by Stx-stimulated cells can amplify the inflammatory processes and the prothrombotic state leading to the constitution of the microangiopathic lesions of HUS. To this day, management of D+HUS involves supportive care mainly based on fluid management, dialysis and red blood cells transfusions. Specific therapies used in D+HUS (plasma infusion, antithrombotic and anti inflammatory agents) failed to improve the course of D+HUS. The use of antibiotics remains not recommended while meta-analysis clearly showed that the use of bactericidal antibiotics could worse the course of D+HUS. In vitro experimentations highlighted that some classes of antibiotics like fluoroquinolones dramatically increase the production and the release of Stx before bacterial lysis and worsen the outcome of D+HUS in animal models. By contrast, azythromycin, a bacteriostatic antibiotic of the macrolides family blocking the protein synthesis in bacteria, has a strong inhibitory effect on Stx production and release by STEC as well as it inhibits the in vitro growth of STEC strains. In addition, azithromycin is able to inhibit the Stx-induced production of inflammatory cytokines which are considered to be essential for the development of D+HUS. Consistently the use of azithromycin in animal models of D+HUS dramatically improved the survival rate. Preliminary data on humans with D+HUS treated with azithromycin highlighted a lower prevalence of severe gastrointestinal involvement than in control patients. All these data supported the hypothesis that azithromycin should have a beneficial effect on D+HUS and should improve the short and long term outcome and deserves to be formally demonstrated in human with D+HUS.

DETAILED DESCRIPTION:
Hemolytic uremic syndrome (HUS) is defined by the combination of microangiopathic hemolytic anemia, thrombocytopenia and acute renal failure. The underlying lesion is thrombotic microangiopathy (TMA) affecting arteriole and capillary walls, with endothelial cells swelling and detachment and thrombi obstructing vascular lumina. Post- diarrheal HUS (D+HUS) is induced by an infection due to E. coli (STEC) producing a Shiga -like toxin (Stx) which is responsible of TMA. Serotype O157:H7 represents 63-97 % of STEC causing D+HUS. Other serotypes frequently implicated in outbreaks are O26:H11, O103:H2, O111:H8, O145:H28 (Mariani - Kurkdjian P et al, 2001) (Espié et al, 2008).

The D+HUS mainly affects children under 3 years and occurs after a prodromal bloody diarrhea. The onset of HUS surrounds 3 to 5 days after the onset of diarrhea. D+HUS is the leading cause of acute renal failure in children under 5 years (Decludt et al. 2000).

In France, 100 to 120 pediatric cases of D+HUS are reported each year. STEC infection was demonstrated in 85 % of cases. In 50 % of cases, one or more persons of the same family have STEC diarrhea without HUS. The death rate in the acute phase is about 2% and 50% of D+HUS requires dialysis. The predictive factors of a poor outcome are an anuria for more than 8 days a neutrophil count>20000/mm3, a severe bowel disease or central nervous system (CNS) involvement (Scheiring et al. 2008). In 65-80 % of cases, a seemingly ad integrum recovery of renal function was observed within the first year after D + HUS onset. However, D+HUS is responsible for a nephron loss that could lead to hypertension, proteinuria and chronic renal failure in the long term. A study performed on 218 patients undergoing D+HUS in the chidhood, highlighted the presence of renal sequelae in nearly 65 % of them with a median follow-up of nearly 20 years. (Fila et al, submitted).

Classically, humans are infected by contaminated food (minced meat undercooked products, unpasteurized milk and cheese...), by the animal environment (especially cattle) or by transmission from person to person. EHEC virulence is associated with the presence of toxins called Shigatoxins (Stx) and the presence of the eae gene, responsible for damage attachment - clearing in the colon and caecum. Two major types of Shigatoxin, Stx1 and Stx2, and many Stx1 or Stx2 variants were identified: three variants for Stx1 and at least, six variants for Stx2. The determination of different profiles variants Stx is considered as predictive of the severity of STEC infections with progression to HUS, especially Stx2d activated and Stx2c After ingestion of contaminated food, STEC are able to withstand the acidity of the stomach and colonize the digestive tract. Toxins produced by the bacteria go through the intestinal epithelium, join the circulatory system and reach their target organs, mainly kidneys and CNS. Indeed, toxins bind to a specific glycolipid receptor, globotriosylceramide (Gb3) on the surface of endothelial cells of target organs (digestive tract, kidney, CNS, pancreas) driving on the one hand, the release of pro-inflammatory factors (TNF- α, IL6, IL8) involved in the formation of lesions of microangiopathy and leading to apoptosis of the target cells (Hurley et al. 2001) (Thorpe et al, 1999) (Zoja et al.2010).

To this day, management of D+HUS requires only supportive care. All specific therapies (antithrombotic and anti inflammatory agents, specific antibodies against Shigatoxin, plasma transfusion and plasma exchange) did not show efficacy (Scheiring et al. 2008) (Loirat et al. 2012).

Several retrospective and prospective studies suggest that antibiotics increase the risk of HUS by release of Stx during bacterial lysis but also to certain types of antibiotics, increased synthesis of Shiga toxin. The meta-analysis performed by Wang et al on the use of antibiotics in patient with STEC diarrhea and D+HUS highlighted an increased risk of developing D+HUS in patients treated with antibiotics (Wang et al. 2000). A second meta-analysis bringing together 20 studies, that compared the risk of HUS occurrence in patients with STEC diarrhea treated or not with antibiotics, has not concluded (Panos et al. 2006). According to these results, antibiotherapy is actually not recommended for patients with diarrhea EHEC and patients with D+HUS (Scheiring et al. 2008). However, these studies did not distinguish between different classes of antibiotics, bringing together all the bacteriostatic antibiotics as well as bactericidal. But, in vitro studies have clearly shown that certain classes of antibiotics such as quinolones induced the production of Shigatoxin (multiplying production by a factor of 100 for ciprofloxacin) while others had a strong inhibitory action as the azithromycin (Ohara et al. 2002 ) .

Azithromycin, an antibiotic of the macrolide family, binds to the 50S subunit of the bacterial ribosome and inhibits protein synthesis by blocking transpeptidation. This mechanism inhibits the production and the release of Shiga toxin in STEC (Ohara et al. 2002). Studies on animal models of D+HUS (mice, piglet) showed a drastic reduction in mortality. Moreover, in addition to its inhibitory action on the synthesis of Stx, azithromycin has a modulating effect on the inflammatory reaction on the vascular endothelium induced by the Shigatoxin that contribute to thrombotic microangiopathy. Indeed, azithromycin dramatically decreased secretion of IL6, IL1 and TNFα (Gantzhorn et al. 2009) (Ohara et al. 2002) (Zhang Q et al. 2009).

Moreover, a recent work from Amran et al performed in a mouse model of D+HUS highlighted a protective effect of azithromycin on the occurrence of neurological inhibition of inflammatory mechanism induced by Shigatoxin in the vascular endothelium brain and neurons (Amran et al. 2013).

On the human being, the German outbreak of D+HUS in O104H4 helped highlight the importance of an early treatment with azithromycin on the eradication of carriage of the bacteria as well as the eradication of Stx in stool (Nitschke et al. 2012). In addition, preliminary data from a retrospective study of D+HUS in Robert Debré hospital showed a lower incidence of severe digestive tract impairment in patients with D+HUS who received treatment with azithromycin compared to the control group (unpublished data).

The objective of a prospective study on patients with D+HUS treated with azithromycin will be to prove its beneficial effects on renal, hematological, digestive tract and neurological impairment seen in D+HUS and to reduce the potential sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 6 months to 18 years old, residing in France, with a D+HUS according to the definition used by the National Institute for Public Health Surveillance (InVS) :
* Renal impairment with a serum creatinine > 60μmol/l in children less than 2 years old and > 75μmol/l over 2 years old
* AND hemolytic anemia defined by hemoglobin < 10g/dl associated with schizocytes ≥ 2%
* Collection of free and informed consent of the holders of parental authority

Exclusion Criteria:

* Age < 6 months and > 18 years.
* Administration of antibiotics in the 15 days preceding the diagnosis of D+HUS.
* Personal or family history of atypical HUS .
* More than 15 days between the onset of diarrhea and the diagnosis of D+HUS.
* Hypersensitivity to azithromycin, erythromycin, or any macrolide
* patient treated with dihydroergotamine, ergotamine or cisapride
* Severe hepatic impairment
* No affiliation to a social security scheme (beneficiary or legal)
* Pregnancy
* Breastfeeding

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR ) assessed with Schwartz formula 2009 | 1 month
  GFR ( ml/min/1.73m ² ) = 39.1 [ Height (m) / Serum creatinine (mg / dl) ] x 0.516 [ 1.8 / cystatin C ( mg / l) ] 0.294 [ 30/urea (mg / dl ) ] x 0.169 [ 1.099 ] x man [ Height (m) / 1.4 ] .188

SECONDARY OUTCOMES:
Hematologic impairment | 1 month
  Hemolysis time defined by the time between the date of diagnosis of D + HUS and the recovery of a normal platelets level (> 150000/mm3 ) Number of packed red blood cells transfusion required during the initial phase of D+HUS
Digestive tract impairment | 1 month
  Occurrence of pancreatitis (defined by a lipase higher than 3 times the upper limit) Occurrence of severe colitis (severe digestive symptoms with bloody diarrhea and ultrasound or CT diagnosis of colitis) Need for parenteral nutrition for more than 72 hours. If yes, duration of parenteral nutrition. Occurence of hepatitis (defined by a SGPT level higher than 3 times the upper limit)
Neurological involvement | 1 month
  Presence or absence of neurological impairment defined by the presence of impaired consciousness and / or confusion and / or convulsions. In the presence of one or more of these signs, neurological impairment must be documented by the completion of a brain imaging (MRI) and electroencephalogram.
Renal impairment | 1 month
  Dialysis, duration of dialysis, anuria, glomerular filtration rate at 1 month, presence of proteinuria and / or a significant microalbuminuria. Blood pressure assessement (according to the standards defined by the Task Force for the size and age of the patient). Time to return to plasma creatinine level < 60μmol/l if the delay is less than one month
One month Survival | 1 month
  occurrence of death or not at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fila, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Arnaud de Villeneuve Hospital, Montpellier, France